CLINICAL TRIAL: NCT06365047
Title: Clinical Investigation to Measure the Changes in the Oral Environment Resulting From a 12 Weeks Exposure to an Arginine Containing Toothpaste
Brief Title: Dry Mouth Toothpaste Study - Comparing Two Toothpastes With Arginine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004926
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigative Arm- Using an 8% Arginine toothpaste (Experimental): For the study period (12 weeks), subjects in the Investigative Arm will be instructed to brush their teeth with an 8% Arginine toothpaste.
  Interventions: Device: 8% Arginine toothpaste
- Control Arm- a 1000 ppm F toothpaste (Active Comparator): For the study period (12 weeks), subjects in the Control Arm will be instructed to brush their teeth with Control Arm- a 1000 ppm F toothpaste.
  Interventions: Drug: 1000 ppm F toothpaste

INTERVENTIONS:
Device: 8% Arginine toothpaste — Investigative
  Arms: Investigative Arm- Using an 8% Arginine toothpaste
Drug: 1000 ppm F toothpaste — Control
  Arms: Control Arm- a 1000 ppm F toothpaste

SUMMARY:
This is a clinical investigation to measure the changes in the oral environment resulting from a 3 month exposure to an arginine containing toothpaste. This study is a double blind, randomized controlled, parallel design. Seventy (70) male and female subjects who meet the inclusion/exclusion criteria will be enrolled in the study. Following oral health evaluations, subjects will be assigned to the treatment schedule and receive their assigned study product.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers 18- 80 years of age and in general good health.
2. Willing and able to understand and sign the informed consent form.
3. Subjects currently taking at least two medications known to cause xerostomia (dry mouth) as a side effect for the last three months.
4. Be willing to conform to the study protocol and procedures.
5. Polypharmacy subjects must score 4 or more on the VAS scale of 0-10 ("How severe is your dryness right now?").
6. Flow of 5 minutes unstimulated saliva should be below 0.16 ml/min.
7. No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the study examiner.
8. Minimum of 10 teeth

Exclusion Criteria:

1. Subjects unable to understand or unwilling to sign the informed consent form.
2. Medical condition which requires premedication prior to dental visits/procedure.
3. Active disease of the hard or soft oral tissues.
4. History of salivary gland disease such as Sjogren's syndrome, Sarcoidosis, or Head and Neck Radiation Therapy.
5. Use of antibiotics or antimicrobial drugs within 30 days prior to study start.
6. Participation in any other clinical study within 1 week prior to enrollment into this study.
7. Subjects who must receive dental treatment during the study dates.
8. Immunocompromised individuals (HIV, AIDS, immunosuppressive drug therapy).
9. Presence of orthodontic bands.
10. Current smokers (if former smoker, should have stopped at least 1 month prior to Visit 1)
11. Use of pilocarpine or other cholinergic stimulating receptor actives prescribed after study enrollment or whose medication dose increases (stable dose for 3 months).
12. People on hormone therapy
13. Pregnant or lactating subjects.
14. Medical condition which prohibits not eating/drinking or chewing gum for four (4) hours prior to your scheduled visits;
15. Subjects who have an infectious disease and/or other blood borne diseases (Hepatitis series, HIV, tuberculosis).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Salivary pH Impact | 12 weeks
  The objective of this clinical research study is to determine if the use of an Arginine containing toothpaste alters the salivary pH of people with xerostomia.

SECONDARY OUTCOMES:
Measuring the change in the oral microbiome | 12 weeks
  The objective of this clinical research study is to determine if the use of an Arginine containing toothpaste alters the oral microbiome (salivary and whole mouth plaque) of people with xerostomia.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Papas, DMD, PhD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States